CLINICAL TRIAL: NCT06491914
Title: A Phase 3b Single-Arm Study of Aflibercept 8 mg in Participants With Neovascular Age-Related Macular Degeneration (nAMD) or Diabetic Macular Edema (DME)
Brief Title: A Phase 3b, Single-Arm Study of Aflibercept 8 mg Dosed Every 4 Weeks in Adult Participants With Neovascular Age-Related Macular Degeneration (nAMD) or Diabetic Macular Edema (DME)
Acronym: ELARA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFTe-HD-OD-2444
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Neovascular Age-Related Macular Degeneration; Diabetic Macular Edema
MeSH Terms: interventions — aflibercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Aflibercept 8 mg (Experimental): Participants previously treated with anti-vascular endothelial growth factor (anti-VEGF) medications
  Interventions: Drug: Aflibercept 8 mg

INTERVENTIONS:
Drug: Aflibercept 8 mg — Administered by intravitreal (IVT) injection
  Other Names: EYLEA®HD; BAY86-5321

SUMMARY:
This study is researching aflibercept high dose (HD), referred to as "study drug", with an experimental dosing regimen. The study is focused on participants with nAMD and DME that have been previously treated with anti-vascular endothelial growth factor (anti-VEGF) medications.

The aim of the study is to see how safe and effective aflibercept HD injections are when given as frequently as every 4 weeks. The study is also looking at what side effects may happen from taking the study drug.

ELIGIBILITY:
Key Inclusion Criteria for Participants with nAMD:

1. ≥50 years of age
2. History of choroidal neovascularization (CNV) lesions secondary to nAMD in the eye study, requiring continued anti-VEGF treatment, as determined by the investigator.

   Key Inclusion Criteria for Participants with DME:
3. ≥18 years of age
4. History of DME with central involvement (in the central subfield on Spectral domain optical coherence tomography [SD-OCT]) in the study eye, requiring continued anti-VEGF treatment, as determined by the investigator

   Key Inclusion for All Participants:
5. Previously treated with ≥3 anti-VEGF IVT injections in the study eye in the 5 months (~150 days) prior to visit 1

Key Exclusion Criteria for Participants with nAMD:

1. Evidence of CNV due to any cause other than nAMD in either eye

   Key Exclusion Criteria for Participants with DME:
2. Evidence of macular edema due to any other cause other than diabetes mellitus in the study eye
3. Active proliferative diabetic retinopathy (DR) in the study eye

NOTE: Other protocol defined inclusion / exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1118 (Actual)
Dates: Start 2024-07-24 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2027-01-07 (Estimated)

PRIMARY OUTCOMES:
Occurrence of treatment-emergent adverse events (TEAEs) | Through week 24
Occurrence of serious TEAEs | Through week 24

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (54):
- United States (53):
  - Win Retina - Arcadia, Arcadia, California
  - California Retina Consultants, Bakersfield, California
  - Retina Specialists of Beverly Hills, Beverly Hills, California
  - Salehi Retina Institute dba Retina Associates of Southern California, Huntington Beach, California
  - South Coast Retina Center, Long Beach, California
  - California Eye Specialists Medical Group, Inc., Pasadena, California
  - Retina Consultants of Southern California, Redlands, California
  - Vrmg Inc, Sacramento, California
  - Retina Consultants of Southern Colorado, Colorado Springs, Colorado
  - Eye care Center of Northern Colorado doing business as Advanced Vision Research Institute, Longmont, Colorado
  - Retina Group of New England, Waterford, Connecticut
  - Advanced Research, LLC, Deerfield Beach, Florida
  - Florida Retina Institute - Jacksonville, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Florida Retina Institute - Orlando, Orlando, Florida
  - Retina Speciality Institute - Pensacola, Florida, Pensacola, Florida
  - Eye Associates of Pinellas, Pinellas Park, Florida
  - Retina Vitreous Associates of Florida Saint Petersburg, St. Petersburg, Florida
  - Retina Vitreous Associates of Florida, Tampa, Florida
  - Center for Retina and Macular Disease, Winter Haven, Florida
  - Georgia Retina, Marietta, Georgia
  - Retina Consultants of Hawaii, Inc., ‘Aiea, Hawaii
  - University Retina and Macula Associates PC - Lemont, Lemont, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Cumberland Valley Retina Consultants-Ophthalmology, Hagerstown, Maryland
  - Mid Atlantic Retina Specialists Hagerstown, Hagerstown, Maryland
  - Opthalmic Consultants of Boston, Boston, Massachusetts
  - Retina Consultants of Minnesota, Edina, Minnesota
  - Deep Blue Retina Clinical Research PLLC, Southaven, Mississippi
  - Vision Research Center Eye Associates of New Mexico, Albuquerque, New Mexico
  - Vitreoretinal Consultants of NY - Westbury, Westbury, New York
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Retina Associates of Cleveland - Beachwood, Beachwood, Ohio
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Tulsa Retina Consultants, Tulsa, Oklahoma
  - EyeHealth Northwest, Portland, Oregon
  - Mid Atlantic Retina, Bethlehem, Pennsylvania
  - Sewickley Eye Group, Sewickley, Pennsylvania
  - Charleston Neuroscience Institute LLC, Ladson, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Tennessee Retina, PC, Nashville, Tennessee
  - Retina Research Institute of Texas, Abilene, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Consultants of Texas, Beaumont, Texas
  - Retina Consultants of Texas - Houston, Bellaire, Texas
  - Texas Retina Associates - Dallas, Dallas, Texas
  - Southwest Retina Consultants, El Paso, Texas
  - Retina Consultants of Texas, Katy, Texas
  - Austin Retina Associates, Round Rock, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas Brown Retina Institute, San Antonio, Texas
  - Retina Consultants Texas, The Woodlands, Texas
  - Pacific Northwest Retina, Bellevue, Washington
- Emanuelli Research and Development Center, Arecibo, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has:
  * received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication or has globally discontinued developed of the product for all indications on or after April 2020 and has no plans for future development
  * made results publicly available (e.g., scientific publication, scientific conference, clinical trial registry)
  * the legal authority to share the data, and
  * ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/